CLINICAL TRIAL: NCT00764153
Title: Hemiarthroplasty or Internal Fixation for Displaced Femoral Neck Fractures - 5 Years Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-2005-OS-2
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Femoral Neck Fractures
Keywords: Displaced Femoral Neck Fractures; Treatment; Function; Pain; Quality of life; Complications; Reoperations; Internal Fixation; Hemiarthroplasty; Activities of Daily Living
MeSH Terms: conditions — Femoral Neck Fractures; Pain | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internal fixation (Other): Closed reduction and internal fixation with two parallel screws (Olmed)
  Interventions: Procedure: Internal fixation
- Bipolar hemiarthroplasty (Other): Hemiarthroplasty with Charnley/ Hastings prosthesis
  Interventions: Procedure: Bipolar hemiarthroplasty

INTERVENTIONS:
Procedure: Bipolar hemiarthroplasty — Lateral approach. FWB.
  Other Names: Charnley/Hastings
  Arms: Bipolar hemiarthroplasty
Procedure: Internal fixation — Fluoroscopic Control. Percutaneous. FWB. Two parallel screws (Olmed)
  Other Names: Olmed (DePuy)
  Arms: Internal fixation

SUMMARY:
An estimated 1.6 million patients sustain a hip fracture every year, about half of these are intracapsular femoral neck fractures. A femoral neck fracture is a life changing event for any patient, and the risk of disability, increased dependence and death is substantial. The main treatment options for displaced femoral neck fractures are internal fixation and arthroplasty. It is established that there are more complications and reoperations after internal fixation, and better short term clinical results with arthroplasty, but knowledge about long term results is lacking.

DETAILED DESCRIPTION:
Patients were included from 2002-2004. Two years follow up was finished by 2006. Patients with displaced intracapsular femoral neck fractures were included and randomized by means of closed numbered envelopes to operation groups:

1. Two parallel screws (Olmed).
2. Hemiarthroplasty with Charnley/ Hastings prosthesis.

A priori one would expect that there would be less morbidity and mortality with the less extensive and quicker operation with parallel screw and that a faster and better rehabilitation would be achieved with hemiarthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Age 60 or above
* Able to walk (any aids allowed)

Exclusion Criteria:

* Anesthesiologically unfit for arthroplasty surgery
* Previous symptomatic hip pathology (i.e. arthritis)
* Pathological fracture
* Delay of more than 96 hours from injury to treatment
* Not living in hospital area

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2002-10; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 5-6 years

SECONDARY OUTCOMES:
Eq-5d | 5-6 years
Barthel Index | 5-6 years
Reoperations and complications | 5-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Madsen, MD PhD, Study Chair — Orthopedic Center, Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Background] Frihagen F, Nordsletten L, Madsen JE. Hemiarthroplasty or internal fixation for intracapsular displaced femoral neck fractures: randomised controlled trial. BMJ. 2007 Dec 15;335(7632):1251-4. doi: 10.1136/bmj.39399.456551.25. Epub 2007 Dec 4. PMID 18056740
- [Background] Frihagen F, Grotle M, Madsen JE, Wyller TB, Mowinckel P, Nordsletten L. Outcome after femoral neck fractures: a comparison of Harris Hip Score, Eq-5d and Barthel Index. Injury. 2008 Oct;39(10):1147-56. doi: 10.1016/j.injury.2008.03.027. Epub 2008 Jul 25. PMID 18656868
- [Background] Stoen RO, Lofthus CM, Nordsletten L, Madsen JE, Frihagen F. Randomized trial of hemiarthroplasty versus internal fixation for femoral neck fractures: no differences at 6 years. Clin Orthop Relat Res. 2014 Jan;472(1):360-7. doi: 10.1007/s11999-013-3245-7. Epub 2013 Aug 24. PMID 23975250